CLINICAL TRIAL: NCT02590744
Title: Effects of Preoperative Using of Eye Patches on Prevention of Preschool Children Emergence Agitation After Cataract Surgery: A Single Center, Prospective, Randomized, Controlled Study.
Brief Title: Effects of Preoperative Using of Eye Patches on Prevention of Emergence Agitation After Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaoliang Gan (Other)
Responsible Party: Sponsor-Investigator, Xiaoliang Gan, associate chief physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Xiaoliang-Gan-2015
Record Dates: First submitted 2015-10-22; First posted 2015-10-29 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Agitation; Child; Anesthesia
Keywords: Emergence Agitation; eye patch; preschool children
MeSH Terms: conditions — Psychomotor Agitation; Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- eye patch (Experimental): cover the sick eye with eye patch for 3 hours preoperatively.
  Interventions: Behavioral: eye patch
- non-eye patch (Placebo Comparator): do not cover the sick eye before surgery.
  Interventions: Behavioral: non-eye patch

INTERVENTIONS:
Behavioral: eye patch — cover the sick eye with eye patch preoperatively for 3 hours
  Other Names: eye shade; eye shield
  Arms: eye patch
Behavioral: non-eye patch — do not cover the sick eye with eye patch preoperatively
  Other Names: eye shade; eye shield
  Arms: non-eye patch

SUMMARY:
This study is a single-center, prospective, randomized, controlled trial. To investigate if preoperative using of eye patch will decrease emergence agitation, and to provide a better method of decreasing emergence agitation to pediatric ophthalmic anesthesiologists.

DETAILED DESCRIPTION:
This study is a single-center, prospective, randomized, controlled trial. To investigate whether preoperative using of eye patches will decrease emergence agitation or not, and to provide a better method of decreasing emergence agitation to pediatric ophthalmic anesthesiologists. The investigators will recruit 180 children undergoing elective cataract surgery, divided into 2 groups by random method. experimental group will cover the effected eye for 3 hours before the operation, while the control group will not. Then the investigators will observe and mesure the incidence of emergence aditation in each group, to assess whether preoperative patch shading can reduce the incidence of postoperative agitation.

ELIGIBILITY:
Inclusion Criteria:

1. Preschool patients undergo elective cataract surgery, whose age are 3 to 7 years.
2. Patients' parents agree to participate in the trial, and sigh the informed consent.

Exclusion Criteria:

1. Patient who can not communicate with medical workers preoperatively.
2. Both of patient's eyes are covered postoperatively.
3. Patient's parents refuse to sign informed consent.
4. The investigators do not think such patient is suitable for our research
5. The patient has serious arrhythmia, abnormal cardiac defect.
6. The patient has suffered from pneumonia, asthma symptoms, bronchitis, or upper respiratory tract infection recent two weeks.
7. The patient has serious disease of the nervous system.
8. The patient has the allergic history of any drug involved in this clinical trial.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
the Padiatric Anesthesia Emergence Agitation Scale | every ten minutes postoperatively, up to 1 hour. Start measuring since the end of surgery until the patient back to ward from postanesthesia care unit.
  measure patients with the pediatric anesthesia emergence agitation scale,the score more than 10 is defined as emergence agitation.

SECONDARY OUTCOMES:
induction compliance checklist | 1 minute before general anesthesia began.
  measure patients with induction compliance checklist before anesthesia.
heart rate (HR) | every ten minutes postoperatively, up to 1 hour. Start measuring since every ten minutes postoperatively, up to 1 hour. Start measuring since the end of surgery until the patient back to ward from postanesthesia care unit.
  measure patients' HR when patient arrived at the post operative care unit
respiration rate(RR) | every ten minutes postoperatively, up to 1 hour. Start measuring since the end of surgery until the patient back to ward from postanesthesia care unit.
  measure patients' RR and SpO2 when patient arrived at the post operative care unit
oxygen saturation(SpO2) | every ten minutes postoperatively, up to 1 hour. Start measuring since the end of surgery until the patient back to ward from postanesthesia care unit.
  measure patients' SpO2 when patient arrived at the post operative care unit
incidence rate of emergence agitation | every ten minutes postoperatively, up to 1 hour. Start measuring since the end of surgery until the patient back to ward from postanesthesia care unit.
  calculate the number of occurrence of emergence agitation

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, PhD, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan ophthalmic center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Lin Y, Shen W, Liu Y, Wang Q, Chen Q, Fang Z, Chi W, Gan X, Liu YZ. Visual preconditioning reduces emergence delirium in children undergoing ophthalmic surgery: a randomised controlled trial. Br J Anaesth. 2018 Aug;121(2):476-482. doi: 10.1016/j.bja.2018.03.033. Epub 2018 May 25. PMID 30032888